CLINICAL TRIAL: NCT03958903
Title: Investigations of Amygdala Function Using Neurophysiological Recording and Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Mahendra Bhati, Clinical Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 42227; DP1MH116506 (NIH); FY18 small grant fund award (Other: Department of Psychiatry, Stanford University)
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Fear; PTSD; Panic Disorder
Keywords: Responsive neurostimulation; Amygdala electrophysiology; Neuropace RNS; Temporal lobe epilepsy; closed-loop brain stimulation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Panic Disorder; Epilepsy, Temporal Lobe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neurophysiological recording and stimulation of amygdala (Experimental): Recording and stimulation of amygdala using Neuropace RNS devices at certain points through out the behavioral tasks.
  Interventions: Device: Amygdala recording and stimulation using Neuropace RNS; Behavioral: Behavioral tasks

INTERVENTIONS:
Device: Amygdala recording and stimulation using Neuropace RNS — Subjects will undergo a series of different, fear-related, behavioral tasks while undergoing amygdala electrophysiology recording and stimulation using the Neuropace RNS devices.
Behavioral: Behavioral tasks — Subjects perform a set of fear related behavioral tasks over 2 days, with 3 tasks each day.In addition to amygdala RNS recording and stimulation, recording of electroencephalography (EEG), electromyography (EMG), and electrodermal activity (EDA) will be performed using standard techniques to capture and quantify the fear response across all tasks.

SUMMARY:
This study aims to specifically examine the in vivo electrophysiology and effects of direct stimulation of the human amygdala during conditioned and evoked fear. Investigators will also examine amygdala electrophysiology and the effects of stimulation during tasks to examine the effects of reward on fear memory.

This study will recruit subjects with a history of temporal lobe epilepsy (TLE) who have undergone neurosurgical implantation with FDA-approved, NeuroPace RNS devices for treatment of seizures. These patients provide a unique cohort with (Responsive Neurostimulation) RNS devices capable of both recording and stimulating the amygdala during performance of fear-based, behavioral tasks.

ELIGIBILITY:
Inclusion Criteria:

* be between age 18-65 years of age
* participants must have received the Neuropace RNS implant to treat their seizures
* have comprehension of instructions in the English language
* be on a stable dose of medications for their epilepsy
* have received the RNS System for Temporal Lobe Epilepsy
* have capacity to provide informed consent

Exclusion Criteria:

* significant cognitive impairment (Mini Mental Status Examination score of less than 20)
* DSM-V diagnosis of alcohol/substance abuse (except nicotine) within the last month or a diagnosis of alcohol/substance dependence (except nicotine) within the last 6 months
* Unable to apply EEG cap
* History of traumatic brain injury
* Active or high suicide risk
* Unable to come to study site/lack of stable housing
* is pregnant or nursing
* Patient's treating neurologist determines that the patient's epilepsy is not stable enough to participate in this study
* Any condition (including psychiatric) which in the judgment of the Investigator would prevent the subject from completion of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
EEG(electroencephalography) amplitude changes | 2 days
  Analyze change in amplitude in microvolts -in resting state EEG recording and EEG recording across all the tasks as determined clinically by the Investigator.
  Investigators will be analyzing stimulus-induced electrophysiological recordings, focusing on Event-Related Potentials (ERPs).
EEG(electroencephalography) frequency changes | 2 days
  Analyze changes in frequency in Hertz- in resting state EEG recording and EEG recording across all the tasks as determined clinically by the Investigator.
  Investigators will be analyzing stimulus-induced electrophysiological recordings, focusing on Event-Related Spectral Potentials (ERSP).
ECoG (ElectroCorticoGraphy) amplitude changes | 2 days
  Quantify changes in ECoG measures as determined clinically by the Investigator.- using intracranial recordings from the Neuropace devices.
  Analyze changes in ECoG amplitude- in resting state and ECoG throughout task and stimulation.
ECoG (ElectroCorticoGraphy) frequency changes | 2 days
  Quantify changes in ECoG measures as determined clinically by the Investigator using intracranial recordings from the Neuropace devices.
  Analyze changes in ECoG frequency - in resting state and ECoG throughout task and stimulation

SECONDARY OUTCOMES:
Electrophysiological changes in EMG | 2 days
  Analyze changes in amplitude of electromyography (EMG) from resting state to EMG recordings across all tasks.
Electrophysiological changes in EDA | 2 days
  Analyze changes in amplitude of electrodermal activity (EDA) from resting state to EMG recordings across all tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Mahendra Bhati, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gross CT, Canteras NS. The many paths to fear. Nat Rev Neurosci. 2012 Sep;13(9):651-8. doi: 10.1038/nrn3301. Epub 2012 Aug 1. PMID 22850830
- [Background] Etkin A, Wager TD. Functional neuroimaging of anxiety: a meta-analysis of emotional processing in PTSD, social anxiety disorder, and specific phobia. Am J Psychiatry. 2007 Oct;164(10):1476-88. doi: 10.1176/appi.ajp.2007.07030504. PMID 17898336
- [Background] Morrell MJ, Halpern C. Responsive Direct Brain Stimulation for Epilepsy. Neurosurg Clin N Am. 2016 Jan;27(1):111-21. doi: 10.1016/j.nec.2015.08.012. PMID 26615113
- [Background] Sato W, Kochiyama T, Uono S, Matsuda K, Usui K, Inoue Y, Toichi M. Rapid amygdala gamma oscillations in response to fearful facial expressions. Neuropsychologia. 2011 Mar;49(4):612-7. doi: 10.1016/j.neuropsychologia.2010.12.025. Epub 2010 Dec 21. PMID 21182851
- [Background] Langevin JP, Koek RJ, Schwartz HN, Chen JWY, Sultzer DL, Mandelkern MA, Kulick AD, Krahl SE. Deep Brain Stimulation of the Basolateral Amygdala for Treatment-Refractory Posttraumatic Stress Disorder. Biol Psychiatry. 2016 May 15;79(10):e82-e84. doi: 10.1016/j.biopsych.2015.09.003. Epub 2015 Sep 11. No abstract available. PMID 26475671
- [Background] Clarke HF, Horst NK, Roberts AC. Regional inactivations of primate ventral prefrontal cortex reveal two distinct mechanisms underlying negative bias in decision making. Proc Natl Acad Sci U S A. 2015 Mar 31;112(13):4176-81. doi: 10.1073/pnas.1422440112. Epub 2015 Mar 16. PMID 25775597

DOCUMENTS (1):
  • Informed Consent Form (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/03/NCT03958903/ICF_000.pdf